CLINICAL TRIAL: NCT07362472
Title: Comparison of Efficacy of Erector Spinae Plane Block Vs Combined Serratus Anterior Plane Block and Pecto-intercostal Fascial Plane Block in Patients Undergoing Breast Cancer Surgery
Brief Title: Comparison of Efficacy of Regional Blocks in Breast Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-23-11
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pain Score; Morphine Consumption
Keywords: Breast surgeries; Erecter spinae plane; serratous anterior plane

STUDY DESIGN:
Intervention Model Description: double blinded randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Interventional regional blocks were provided by consultants with privileges of nerve blocks. Patients, investigators and nursing staff accessing pain score were blinded from the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erecter spinae plane block (Active Comparator): Ultrasound guided 30ml erecter spinae plane block was provided with standard bupivacaine (2mg/kg)
  Interventions: Procedure: Regional nerve blocks
- serratous anterior plane block and pecto-intercoastal facial plane block (Active Comparator): Ultrasound guided 30ml serratous anterior plane block and pecto-intercoastal facial plane block was provided with standard bupivacaine (2mg/kg)
  Interventions: Procedure: Regional nerve blocks

INTERVENTIONS:
Procedure: Regional nerve blocks — In these interventions we compared two regional blocks (serratous anterior & pecto intercoastal facial plane block) techniques vs one regional block (erecter spinae plane block)

SUMMARY:
After Standardized anesthetic induction patients were randomly given regional blocks. Group A recieved erecter spinae plane block & group B recieved combined serratous anterior and pecto-intercoatal facial plane block. Their mean morphine consumption were followed for the next 24 hours.

DETAILED DESCRIPTION:
Subjects who are fulfilling the inclusion criteria will be included in the study after taking informed consent once approved by scientific review committee and Institutional review board.Subjects will be randomly divided into two groups by using a computer generated table using website Research Randomizer which will allocate the subjects randomly in two groups.Non probability consecutive sampling technique will used.Day cases are not included and major breast surgeries with post operative admission are included in study.Procedure will be done by the consultant having privilege to perform the block.Group A will be receiving ultrasound guided Erector spinae plane block before surgical incision with bupivacaine (maximum dose 2mg/kg) having total volume of 30ml. Group B will receive ultrasound guided combined serratus anterior plane block( in which local anesthetic is injected between the serratus anterior and latissimus dorsi muscles at level of 5th rib in mid to posterior axillary line)and pecto-intercostal plane block(in which local anesthetic is injected between the pectoral and intercostal muscle layer in 4th rib pecto-sternal region)before surgical procedure with same dose of bupivacaine (maximum dose 2mg/kg) with total volume of 30ml.Induction of anesthesia will be done before block using 2-3mg/kg Propofol, 0.5mg/kg Atracurium and placement of supraglottic airway device will be done in each group as part of standardization(5). Maintenance of anesthesia will be done with inhalational Sevoflurane, oxygen and air mixture. Every patient will be given Paracetamol 1g and Diclofenac 75mg for analgesia and dexamethasone 8mg if not contraindicated intraoperatively. Rescue analgesia with 0.05-0.1mg/kg Morphine will be administered intraoperatively in a titrated fashion to all those patients for pain with 20% increase in Heart rate and blood pressure from base line.Ondansetron(0.1mg/kg) IV as antiemetic and neostigmine/glycopyrrolate as a reversal agent will be used.Pain score will be assessed by RN registered nurse during first hour post operatively, at discharge from PACU using Numeric Rating Scale(NRS)and at 24 hours postoperatively on IPD using NRS and will be recorded in electronic record system of hospital. Any patient with a score of more than 3 will be administered IV morphine (0.1mg/kg). Post operative analgesic plan is multimodal with Paracetamol (1gm IV TID) and IV diclofenac 50mg BID (if no contraindication) along with opioid on PRN basis. All data will be recorded on a Performa from electronic record system (attached at the end).

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing major breast cancer surgeries (modified radical mastectomy, breast reconstruction with implants).
* American society of anesthesiologist Grade 1 & 2
* Age between 18 to 45 years

Exclusion Criteria:

* Patient's refusal
* Emergency cases
* Patients having uncontrolled diseases like asthma, COPD or other lung diseases
* History of allergy from the drugs being used during the study
* Pregnant patients
* Patients with coagulopathies/bleeding disorders
* Patients undergoing bilateral major breast cancer surgery.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Breast cancer surgeries
Enrollment: 60 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
mean morphine consumption | 24 hours
  We calculated and compared mean morphine consumption in first 24 hours post operatively among the 2 groups.

SECONDARY OUTCOMES:
Pain score | 24 hours
  We accessed pain scores post operatively in PACU at regular intervals and later on in inpatient for first 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hamood Ur Rehman, MBBS, Principal Investigator — Shaukat Khanam Memorial Cancer Hospital & Research Centre Lahore
Locations (1):
- Shaukat Khanam Memorial Cancer Hospital & Research Centre Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finnerty DT, McMahon A, McNamara JR, Hartigan SD, Griffin M, Buggy DJ. Comparing erector spinae plane block with serratus anterior plane block for minimally invasive thoracic surgery: a randomised clinical trial. Br J Anaesth. 2020 Nov;125(5):802-810. doi: 10.1016/j.bja.2020.06.020. Epub 2020 Jul 11. PMID 32660716